CLINICAL TRIAL: NCT02528708
Title: A Program to Evaluate Riastap® and FIBTEM® for the Early Control and Treatment of Postpartum Hemorrhage (PERFECT PPH)
Acronym: PERFECT PPH
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study never began.
Sponsor: Yale University (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1504015615
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Postpartum Hemorrhage
Keywords: fibrinogen concentrate; coagulation
MeSH Terms: conditions — Postpartum Hemorrhage; Thrombosis | interventions — Fibrinogen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): At the same time of randomization code generation, blood samples for a baseline ROTEM® analysis will be drawn, and blood products will be ordered. Patients will be eligible to receive study drug (fibrinogen concentrate or 0.9% saline solution), according to the randomization code previously generated, only if FIBTEM® - A10 value is <18 mm (corresponding to a MCF value of <20 mm, that is a plasma fibrinogen level <3 g/L).
  Interventions: Drug: Placebo
- Fibrinogen concentrate (Experimental): At the same time of randomization code generation, blood samples for a baseline ROTEM® analysis will be drawn, and blood products will be ordered. Patients will be eligible to receive study drug (fibrinogen concentrate or 0.9% saline solution), according to the randomization code previously generated, only if FIBTEM® - A10 value is <18 mm (corresponding to a MCF value of <20 mm, that is a plasma fibrinogen level <3 g/L).
  Interventions: Drug: fibrinogen concentrate

INTERVENTIONS:
Drug: fibrinogen concentrate — The dose of fibrinogen concentrate needed to achieve this target will be calculated using a formula that accounts for the baseline FIBTEM® - A10 value and the patient's body weight assessed at hospital admission . In general, a 70-kg patient requires a fibrinogen dose of approximately 0.5 g to increase the MCF by approximately 1 mm.
  Other Names: Riastap
  Arms: Fibrinogen concentrate
Drug: Placebo — 0.9% saline solution
  Other Names: saline
  Arms: Placebo

SUMMARY:
In this prospective, single-center, randomized, placebo-controlled, double-blind clinical trial, parturients with primary PPH are eligible for treatment with fibrinogen concentrate following both vaginal delivery and cesarean section complicated by an estimated blood loss (EBL) >1000 mL and an ongoing bleeding notwithstanding standard treatment measures (volume replacement, uterine massage, and uterotonic agents).

DETAILED DESCRIPTION:
The proposed trial targets early detection and treatment of fibrinogen depletion in PPH. A widespread belief in the benefits of early fibrinogen substitution in cases of PPH has led to an increased use for this indication. The PERFECT PPH aims to provide an evidence-based knowledge for the recommendation of the early use of fibrinogen concentrate in PPH.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from participant
* Age ≥18 years and <50 years
* Primary PPH defined as bleeding from uterus and/or the birth canal within 24 hours postpartum
* Vaginal delivery or Cesarean delivery (irrespective of etiology of PPH, such as accreta), with EBL >1000 mL and ongoing bleeding notwithstanding standard treatment measures (volume replacement, uterine massage, uterotonic agents)
* FIBTEM®- A10 <18 mm (corresponding to a MCF value of <20 mm and to a plasma fibrinogen level approximately <3 g/L)

Exclusion Criteria:

* Refusal to give written informed consent
* Refusal to receive blood transfusion
* Known inherited deficiencies of coagulation
* Personal history of thrombosis
* Either pre-pregnancy or ante-partum antithrombotic treatment due to increased risk of thrombosis
* Administration of Platelets, FFP or cryotherapy prior to study drug

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
maximum clot firmness (MCF via FIBTEM A10) | 15 minutes
  fib-tem® is a ready-to-use ROTEM® system reagent for use with citrated whole blood. It assesses the clot firmness of the fibrin clot. This is influenced mainly by the fibrinogen- and F XIII levels of the blood sample and by fibrin polymerisation disorders. The reagent contains a powerful platelet inhibitor; therefore only a fibrin clot is formed and measured. MCF is measured as the maximal amplitude of the curve.
maximum clot firmness (MCF via FIBTEM A10) | 1 hour
  fib-tem® is a ready-to-use ROTEM® system reagent for use with citrated whole blood. It assesses the clot firmness of the fibrin clot. This is influenced mainly by the fibrinogen- and F XIII levels of the blood sample and by fibrin polymerisation disorders. The reagent contains a powerful platelet inhibitor; therefore only a fibrin clot is formed and measured. MCF is measured as the maximal amplitude of the curve.
maximum clot firmness (MCF via FIBTEM A10) | 6 hours
  fib-tem® is a ready-to-use ROTEM® system reagent for use with citrated whole blood. It assesses the clot firmness of the fibrin clot. This is influenced mainly by the fibrinogen- and F XIII levels of the blood sample and by fibrin polymerisation disorders. The reagent contains a powerful platelet inhibitor; therefore only a fibrin clot is formed and measured. MCF is measured as the maximal amplitude of the curve.
maximum clot firmness (MCF via FIBTEM A10) | 24 hours
  fib-tem® is a ready-to-use ROTEM® system reagent for use with citrated whole blood. It assesses the clot firmness of the fibrin clot. This is influenced mainly by the fibrinogen- and F XIII levels of the blood sample and by fibrin polymerisation disorders. The reagent contains a powerful platelet inhibitor; therefore only a fibrin clot is formed and measured. MCF is measured as the maximal amplitude of the curve.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Paidas, MD, Principal Investigator — Yale University